CLINICAL TRIAL: NCT03181048
Title: Single-Blind Randomized Clinical Trial of Concomitant Hip Arthroscopy During Periacetabular Osteotomy for the Management of Hip Dysplasia
Brief Title: Clinical Trial of Concomitant Hip Arthroscopy During PAO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rafael J. Sierra, M.D., Professor of Orthopedics, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-001014
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Hip Dysplasia
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be randomized in a 1:1 fashion. The first arm will be the "PAO alone" group who will receive a standard periacetabular osteotomy (PAO) on the day of surgery. The second arm will be the "PAO + HA" group who will receive a PAO and hip arthroscopy (HA) on the day of surgery. Any pathology if present that can be corrected with the arthroscope (cartilage and labral abnormalities) will be addressed. This will be followed by a standard PAO. Patients from both groups will have dressings placed in the location of hip arthroscopy portals to remain blinded to the treatment arm during the perioperative period. Only patients in the PAO + HA group will have incisions and sutures under these dressings. The dressings will come off for all patients after 2 weeks, which is standard of care. All other study team members will remain unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periacetabular osteotomy (Experimental): Standard periacetabular osteotomy on the day of surgery.
  Interventions: Procedure: Periacetabular osteotomy
- Periacetabular osteotomy with hip arthroscopy (Active Comparator): Hip arthroscopy on the day of surgery, followed by a standard periacetabular osteotomy.
  Interventions: Procedure: Periacetabular osteotomy with hip arthroscopy

INTERVENTIONS:
Procedure: Periacetabular osteotomy — The Bernese periacetabular osteotomy has become the osteotomy of choice in North America for correction of the dysplastic hip. The ability to position the acetabular component in a specifically desired position for each individual patient improves joint biomechanics, restores joint balance and stability, and offloads the structures at risk for damage such as the labrum and the adjacent articular cartilage.
  Arms: Periacetabular osteotomy
Procedure: Periacetabular osteotomy with hip arthroscopy — An intraarticular assessment with hip arthroscopy (HA) at the time of periacetabular osteotomy allows the surgeon to assess and treat the associated labral and chondral pathology and allows the surgeon to treat abnormalities of the femoral head junction.
  Arms: Periacetabular osteotomy with hip arthroscopy

SUMMARY:
The study will assess the outcomes of patients treated with concomitant hip arthroscopy at the time of periacetabular osteotomy (PAO) for patients with hip dysplasia compared with patients treated with PAO alone.

DETAILED DESCRIPTION:
There are currently no absolute indications for intraarticular assessment at the time of periacetabular osteotomy (PAO). Based on investigators' review of the literature and experience, patients who may benefit from intraarticular assessment are those with radiographic or MRI evidence of damage where an intraarticular inspection may help in determining whether a PAO is a reasonable procedure, those with mechanical symptoms likely related to labral pathology, round ligament or cartilage problems and those with hip dysplasia and cam deformities with limited range of motion that may benefit from femoral head neck junction osteochondroplasty. However, despite these relative indications today there is no clear evidence to suggest that these patients will do better than those that do not have intraarticular work done. Hence, the objective of this project is to determine whether intraarticular work at the time of PAO surgery leads to improved pain and function when compared to patients that do not undergo intraarticular work at the time of PAO.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hip dysplasia (DDH) electing periacetabular osteotomy (PAO) for treatment
* Skeletally mature
* Age 15 - 55
* Tonnis Grade 0 or 1 osteoarthritis (minimal or no arthritis)
* Ability to receive a standard of care preoperative (magnetic resonance imaging) MRI arthrogram of the hip

Exclusion Criteria:

* Pregnant women
* Previous surgery about the hip
* Patients receiving PAO for acetabular retroversion in the absence of DDH
* Previous hip arthroscopy to address intra-articular pathology

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Estimated)
Dates: Start 2017-08-23 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Mean score of Hip Disability and Osteoarthritis Outcome (Hoos) | 1 year follow-up time point
  Score ranges from 0-100 with higher scores representing better function.
Mean score of Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 1 year follow-up time point
  The scores range from 0-4 in 24 different categories that are broken up into three subcategories: pain, stiffness and physical function.
Mean score of University California Los Angeles (UCLA) activity assessment | 1 year follow-up time point
  Measured on a 1-10 scale: 1) wholly inactive, dependent on others; 2) mostly inactive, restricted to minimal activities of daily living; 3) sometimes participate in mild activities such as walking, limited housework, or shopping; 4) regularly participate in mild activities; 5) sometimes participate in moderate activities such as swimming and unlimited housework or shopping; 6) regularly participate in moderate activities; 7) regularly participate in active events such as bicycling; 8) regularly participate in very active events such as bowling or golf; 9) sometimes participate in impact sports such as jogging, tennis, or skiing, or heavy labor; and 10) regularly participate in impact sports.
Mean score of the Marx Activity Scale (MARX) | 1 year follow-up time point
  Score is measured from 0-4.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Sierra, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Only study personnel authorized by the investigator will collect data/enroll subjects. Data will be stored in electronic files and/or a cabinet, with access to study personnel as authorized by the investigator. The investigator will review the data on a regular basis (at least annually) to verify the validity of the data.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials